CLINICAL TRIAL: NCT04043494
Title: LBL 2018 - International Cooperative Treatment Protocol for Children and Adolescents With Lymphoblastic Lymphoma
Brief Title: International Cooperative Treatment Protocol for Children and Adolescents With Lymphoblastic Lymphoma
Acronym: LBL 2018
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKM17_0023; 2017-001691-39 (EudraCT Number)
Record Dates: First submitted 2019-07-15; First posted 2019-08-02 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-07

CONDITIONS: Lymphoblastic Lymphoma, Childhood
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Daunorubicin; Doxorubicin; Ifosfamide; Mercaptopurine; Methotrexate; pegaspargase; Prednisone; Prednisolone; Thioguanine; Vincristine; Vindesine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- SR I/II: R1 into protocol Ia-Pred (Other): 1. cytoreductive prephase with prednisone
  2. standard induction phase (protocol Ia-prednisone)
  3. consolidation phase (protocol Ib)
  4. non-HR extra-compartment phase (protocol M)
  5. maintenance therapy
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: PEG asparaginase; Drug: Prednisone; Drug: Prednisolone; Drug: Vincristine
- SR I/II: R1 into protocol Ia-Dexa (Experimental): 1. cytoreductive prephase with prednisone
  2. experimental induction phase (protocol Ia-dexamethasone)
  3. consolidation phase (protocol Ib)
  4. non-HR extra-compartment Phase (protocol M)
  5. maintenance therapy
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Daunorubicin; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: PEG asparaginase; Drug: Prednisone; Drug: Prednisolone; Drug: Vincristine
- SR: R1 into protocol Ia-Pred (Other): 1. cytoreductive prephase with prednisone
  2. standard induction phase (protocol Ia-prednisone)
  3. consolidation phase (protocol Ib)
  4. non-HR extra-compartment phase (protocol M)
  5. reintensification phase (protocol II)
  6. maintenance therapy
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Daunorubicin; Drug: Doxorubicin; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: PEG asparaginase; Drug: Prednisone; Drug: Prednisolone; Drug: Thioguanine; Drug: Vincristine
- SR: R1 into protocol Ia-Dexa (Experimental): 1. cytoreductive prephase with prednisone
  2. experimental induction phase (protocol Ia-dexamethasone)
  3. consolidation phase (protocol Ib)
  4. non-HR extra-compartment phase (protocol M)
  5. reintensification phase (protocol II)
  6. maintenance therapy
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Daunorubicin; Drug: Doxorubicin; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: PEG asparaginase; Drug: Prednisone; Drug: Prednisolone; Drug: Thioguanine; Drug: Vincristine
- HR: R1 into "Pred" and R2 into non-HR extra-compartment phase (Other): 1. cytoreductive prephase with prednisone
  2. standard induction phase (protocol Ia-prednisone)
  3. consolidation phase (protocol Ib)
  4. non-HR extra-compartment phase (protocol M)
  5. reintensification phase (protocol II)
  6. maintenance therapy
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Daunorubicin; Drug: Doxorubicin; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: PEG asparaginase; Drug: Prednisone; Drug: Prednisolone; Drug: Thioguanine; Drug: Vincristine
- HR: R1 into "Dexa" and R2 into non-HR extra-compartment phase (Experimental): 1. cytoreductive prephase with prednisone
  2. experimental induction phase (protocol Ia-dexamethasone)
  3. consolidation phase (protocol Ib)
  4. non-HR extra-compartment phase (protocol M)
  5. reintensification phase (protocol II)
  6. maintenance therapy
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Daunorubicin; Drug: Doxorubicin; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: PEG asparaginase; Drug: Prednisone; Drug: Prednisolone; Drug: Thioguanine; Drug: Vincristine
- HR: R1 into "Pred" and R2 into HR extra-compartment phase (Experimental): 1. cytoreductive prephase with prednisone
  2. standard induction phase (protocol Ia-prednisone)
  3. consolidation phase (protocol Ib*)
  4. HR extra-compartment phase (intensified protocol M)
  5. reintensification phase (protocol II)
  6. maintenance therapy
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Daunorubicin; Drug: Doxorubicin; Drug: Ifosfamide; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: PEG asparaginase; Drug: Prednisone; Drug: Prednisolone; Drug: Thioguanine; Drug: Vincristine; Drug: Vindesine
- HR: R1 into "Dexa" and R2 into HR extra-compartment phase (Experimental): 1. cytoreductive prephase with prednisone
  2. experimental induction phase (protocol Ia-dexamethasone)
  3. consolidation phase (protocol Ib*)
  4. HR extra-compartment phase (intensified protocol M)
  5. reintensification phase (protocol II)
  6. maintenance therapy
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Daunorubicin; Drug: Doxorubicin; Drug: Ifosfamide; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: PEG asparaginase; Drug: Prednisone; Drug: Prednisolone; Drug: Thioguanine; Drug: Vincristine; Drug: Vindesine

INTERVENTIONS:
Drug: Cyclophosphamide — Part of standard chemotherapy and included in the experimental treatment phase protocol Ib* (Randomization 2) and in the experimental treatment phase Intensified Protocol M (Randomization R2)
Drug: Cytarabine — No involvement of CNS: Part of standard chemotherapy and included in the experimental treatment phase protocol Ib* (Randomization 2) and in the experimental treatment phase Intensified Protocol M (Randomization R2).
  Involvement of CNS: Part of standard chemotherapy and included in the experimental treatment phase Protocol Ia-Dexamethasone (Randomization R1), in the experimental treatment phase Protocol Ib* (Randomization R2) and in the experimental treatment phase Intensified Protocol M (Randomization R2)
Drug: Dexamethasone — Part of the experimental therapy in Randomization R1 (Protocol Ia-Dexamethasone) and in Randomization R2 (Intensified Protocol M)
  Arms: HR: R1 into "Dexa" and R2 into HR extra-compartment phase; HR: R1 into "Dexa" and R2 into non-HR extra-compartment phase; HR: R1 into "Pred" and R2 into HR extra-compartment phase; HR: R1 into "Pred" and R2 into non-HR extra-compartment phase; SR I/II: R1 into protocol Ia-Dexa; SR: R1 into protocol Ia-Dexa; SR: R1 into protocol Ia-Pred
Drug: Daunorubicin — Part of standard chemotherapy and included in the experimental treatment phase Protocol Ia-Dexamethasone (Randomization R1), in the experimental treatment phase Protocol Ib* (Randomization R2) and in the experimental treatment phase Intensified Protocol M (Randomization R2)
Drug: Doxorubicin — Part of standard chemotherapy
  Arms: HR: R1 into "Dexa" and R2 into HR extra-compartment phase; HR: R1 into "Dexa" and R2 into non-HR extra-compartment phase; HR: R1 into "Pred" and R2 into HR extra-compartment phase; HR: R1 into "Pred" and R2 into non-HR extra-compartment phase; SR: R1 into protocol Ia-Dexa; SR: R1 into protocol Ia-Pred
Drug: Ifosfamide — Part of the experimental therapy in Randomization R2 (Intensified Protocol M)
  Arms: HR: R1 into "Dexa" and R2 into HR extra-compartment phase; HR: R1 into "Pred" and R2 into HR extra-compartment phase
Drug: 6-Mercaptopurine — Part of standard chemotherapy and included in the experimental treatment phase protocol Ib* (Randomization 2) and in the experimental treatment phase Intensified Protocol M (Randomization R2)
Drug: Methotrexate — Part of standard chemotherapy and included in the experimental treatment phase Protocol Ia-Dexamethasone (Randomization R1), in the experimental treatment phase Protocol Ib* (Randomization R2) and in the experimental treatment phase Intensified Protocol M (Randomization R2)
Drug: PEG asparaginase — Part of standard chemotherapy and included in the experimental treatment phase Protocol Ia-Dexamethasone (Randomization R1) and in the experimental treatment phase Protocol Ib* (Randomization R2)
Drug: Prednisone — Part of standard chemotherapy
Drug: Prednisolone — No involvement of CNS: Part of standard chemotherapy. Involvement of CNS: Part of standard chemotherapy and included in the experimental treatment phase Protocol Ia-Dexamethasone (Randomization R1), in the experimental treatment phase Protocol Ib* (Randomization R2) and in the experimental treatment phase Intensified Protocol M (Randomization R2
Drug: Thioguanine — Part of standard chemotherapy
  Arms: HR: R1 into "Dexa" and R2 into HR extra-compartment phase; HR: R1 into "Dexa" and R2 into non-HR extra-compartment phase; HR: R1 into "Pred" and R2 into HR extra-compartment phase; HR: R1 into "Pred" and R2 into non-HR extra-compartment phase; SR: R1 into protocol Ia-Dexa; SR: R1 into protocol Ia-Pred
Drug: Vincristine — Part of standard chemotherapy and included in the experimental treatment phase Protocol Ia-Dexamethasone (Randomization R1) and in the experimental treatment phase Intensified Protocol M (Randomization R2)
Drug: Vindesine — Part of the experimental therapy in Randomization R2 (Intensified Protocol M)
  Arms: HR: R1 into "Dexa" and R2 into HR extra-compartment phase; HR: R1 into "Pred" and R2 into HR extra-compartment phase

SUMMARY:
Primary objectives:

* Randomization R1, all patients eligible: To examine, whether the cumulative incidence of relapses with involvement of the CNS (CNS relapse, pCICR) can be decreased by a modified induction therapy including dexamethasone (experimental arm) instead of prednisone (standard arm)
* Randomization R2, only patients with high risk LBL eligible: to examine, whether the probability of event-free survival (pEFS) in these patients can be improved by receiving an intensified treatment arm versus a standard treatment arm (as used in the EURO-LB 02)

DETAILED DESCRIPTION:
The trial LBL 2018 is a collaborative prospective, multi-national, multi-center, randomized clinical trial for the treatment of children and adolescents with newly diagnosed lymphoblastic lymphoma.

The LBL 2018 trial will be open for the qualified centers of following participating study Groups (core study cohort): AIEOP (Italy), BFM (Austria, Czech Republic, Germany, Switzerland), BSPHO (Belgium), CoALL (Germany), DCOG (The Netherlands), NOPHO (Denmark, Finland, Norway, Sweden), PPLLSG (Poland), SEHOP (Spain) and SFCE (France). HKPHOSG (Hong Kong), HPOG (Hungary), ISPHO (Israel), NSPHO (Moscow), SHOP (Portugal) and SPS (Slovak Republic) start patient recruitment into the extended study cohort (without randomization). Over the trial period study groups may switch from the extended study cohort to the core study cohort.

Primary objectives:

* Randomization R1, all patients eligible: To examine, whether the cumulative incidence of relapses with involvement of the CNS (CNS relapse, pCICR) can be decreased by a modified induction therapy including dexamethasone (experimental arm) instead of prednisone (standard arm)
* Randomization R2, only patients with high risk LBL eligible: to examine, whether the probability of event-free survival (pEFS) in these patients can be improved by receiving an intensified treatment arm versus a standard treatment arm (as used in the EURO-LB 02)

Patients are stratified into 3 different risk groups according to CNS status, immunophenotype, genetic markers and stage of disease at diagnosis: high risk group (HR), standard risk group I/II (SR I/II) and standard risk group (SR).

Patients in the risk groups SR I/II and SR are randomized (R1) in two arms after a cytoreductive prephase with prednisone. Patients in standard arm receive the standard induction phase with prednisone. Patients in the experimental arm receive an induction phase with dexamethasone instead of prednisone.

In SR group, induction phase is followed by the consolidation phase, the non-HR extra-compartment phase with HD-MTX (high-dose methotrexate), the reintensification phase and the maintenance therapy for the total therapy duration of 24 months. In SR I/II group, patients receive no reintensification phase. The Induction phase is followed by the consolidation phase, the non-HR extra-compartment phase and the maintenance therapy for the total therapy duration of 24 months.

Patients in the HR group are eligible for randomization (R1) as outlined above. In addition high risk patients are eligible for second randomization (R2) at the end of induction phase. In the standard arm, HR-patients receive the consolidation phase and the non-HR extra-compartment phase. In the experimental arm, HR-patients receive a consolidation phase including two additional doses of PEG asparaginase and the HR-intensified extra-compartment phase consisting of two high risk courses alternating with two HD-MTX courses. Either phase is followed by the reintensification phase and the maintenance therapy for the total therapy duration of 24 months.

Patients with involvement of the CNS (CNS positive) are stratified to the high risk group (HR) and are eligible for both randomizations (R1 and R2). Additionally, patients with CNS involvement (CNS positive) receive intensified intrathecal therapy. Intrathecal therapy consists of TIT (triple intrathecal therapy) after diagnosis of CNS involvement. TIT is administered twice weekly until clearance of blasts in the cerebrospinal fluid is achieved. Further intrathecal therapy is provided at the same points of time as for patients without CNS involvement, but TIT instead of MTX IT. In addition, patients receive four additional doses of TIT during maintenance. Cranial irradiation is omitted for patients with CNS involvement.

ELIGIBILITY:
Inclusion criteria:

* newly diagnosed lymphoblastic lymphoma
* age <18 years
* patient enrolled in a participating center
* written informed consent of patient (>14 years of age or according to local law and regulation) and parents to trial participation and transfer and processing of data
* willingness of patients and the investigator/pathologist to provide adequate slides/blocks for reference (molecular) pathology and international pathology panel and/or fresh or fresh frozen samples for genetic risk group stratification if these samples are available after standard diagnostic procedures.

Exclusion criteria:

* lymphoblastic lymphoma as secondary malignancy
* non-lymphoma related relevant medical, psychiatric or social conditions incompatible with trial treatment, including among others

  * prior organ transplant
  * severe immunodeficiency
  * demyelinating Charcot-Marie Tooth syndrome
  * serious acute or chronic infections, such as HIV, VZV and tuberculosis
  * urinary tract infection, cystitis, urinary outflow obstruction, severe renal impairment (creatinine clearance less than 20 ml/min)
  * severe hepatic impairment (bilirubin >3 times ULN, transaminases >10 times ULN)
  * myocardial insufficiency, severe arrhythmias
  * ulcers of the oral cavity and known active gastrointestinal ulcer disease
  * known hypersensitivity to any IMP and to any excipient (listed in section 6.1 of the respective SmPC)
* steroid pre-treatment with ≥ 1 mg/kg/d for more than two weeks during the last month before diagnosis
* vaccination with live vaccines within 2 weeks before start of protocol treatment
* treatment started according to another protocol or pre-treatment with cytostatic drugs
* participation in another clinical trial that interferes with the protocol, except NHL-BFM Registry 2012 and trials with different endpoints, involving aspects of supportive treatment, which can run parallel to LBL 2018 without influencing the outcome of this trial (e.g. trials on antiemetics, antibiotics, strategies for psychosocial support)
* evidence of pregnancy or lactation period
* sexually active adolescents not willing to use highly effective contraceptive method (pearl index < 1) until 12 months after end of cytostatic therapy

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 683 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2027-11-22 (Estimated); Study Completion 2027-11-22 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of relapse with involvement of the CNS (CNS-relapse, pCICR) | through study completion, maximal 7.25 years
  The time to relapse is defined as the time from randomization to the first relapse or the date of last follow-up. Other events (non-response, progressive disease, relapse, second malignancy or death before and in CR) will be taken into account as competing events.
Estimated probability of event-free survival (pEFS) | through study completion, maximal 7.25 years
  The pEFS is defined as the time from randomization to the first event (non-response, progressive disease, relapse, second malignancy or death from any cause) or date of last follow-up.

SECONDARY OUTCOMES:
Survival (pOS) | through study completion, maximal 7.25 years
  Survival (pOS) is defined as time from diagnosis to death due to any cause or to the date of last contact for patients alive
Frequency of treatment-related toxicity overall and in specific protocol elements, randomized arms and during follow up | through study completion, maximal 7.25 years
Frequency of treatment-related mortality overall and in specific protocol elements, randomized arms and during follow up | through study completion, maximal 7.25 years
Frequency of adverse events of interest and severe adverse events overall | through study completion, maximal 7.25 years
Rate of evaluable patients for risk group stratification | during recruitment
Cumulative incidence of relapses in association with molecular markers | through study completion, maximal 7.25 years
Cumulative incidence of relapses in association with minimal residual disease results | through study completion, maximal 7.25 years

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Burkhardt, Prof. Dr. Dr., Principal Investigator — University Hospital Muenster, Klinik für Kinder- und Jugendmedizin - Pädiatrische Hämatologie und Onkologie
Locations (228):
- Austria (5):
  - Univ.Klinik für Kinder- und Jugendheilkunde Graz, Klin. Abteilung für pädiatrische Hämato-Onkologie, Graz
  - Univ.Klinik für Kinder- und Jugendheilkunde Innsbruck, Universitätsklinik für Pädiatrie I, Innsbruck
  - Kepler Universitätsklinikum, Med Campus IV / Onkologie, Linz
  - LKH Salzburg, Universitätsklinik für Kinder- und Jugendheilkunde, Kinderonkologie, Salzburg
  - St. Anna Kinderspital, Vienna
- Belgium (8):
  - Hôpital Universitaire des Enfants Reine Fabiola (ULB), Pédiatrie hémato-oncologie, Brussels
  - University Hospital Brussels, Pediatrische oncologie, Brussels
  - Cliniques Universitaires Saint-Luc (UCL), Hématologie et oncologie pédiatrique, Brussels
  - UZ Antwerpen Kinderhemato-oncologie, Edegem
  - University Hospital Gent Pediatrische hemato-oncologie, Ghent
  - University Hospitals Leuven, Kinderhemato-oncologie, Leuven
  - CHR Citadelle Hémato - oncologie pédiatrique, Liège
  - CHR Citadelle Hémato - oncologie pédiatrique, Montegnée
- Hong Kong Children's Hospital, Hong Kong, China
- Czechia (2):
  - Dept. of Pediatric Oncology, University Hospital Brno and Faculty of Medicine, Masaryk University Cernopolni, Brno
  - Dept. of Pediatric Hematology and Oncology. University Hospital Motol and 2nd Medical School, Charles University, Prague
- Denmark (4):
  - University Hospital Aalborg, Nord, Department of Pediatrics, Aalborg
  - Aarhus University Hospital, Department of Pediatrics, Aarhus
  - Børneonkologisk afsnit 5054, BørneUngeKlinikken, Juliane Marie Centret, Rigshospitalet, Copenhagen
  - H.C. Andersens Children Hospital, Odense University Hospital, Odense
- Finland (5):
  - Helsinki University Hospital, Department of Pediatric Hematology and Oncology, Helsinki
  - Kuopio University Hospital, Department of Pediatric Hematology and Oncology, Kuopio
  - University Hospital of Oulu, Paediatric Haematology and Oncology, Oulu
  - Tampere University Hospital, Paediatric Haematology and Oncology, Tampere
  - Turku University Hospital, Paediatric and Adolescent Haematology and Oncology, Turku
- France (29):
  - Service d'oncolologie, Hématologie pédiatrique. CHU Amiens, Avenue René Laënnec - SALOUEL, Amiens
  - Pôle Femme Mère Enfant ; Unité d'Hématologie/Oncologie pédiatrique, CHU Angers, Angers
  - Hématologie Oncologie pédiatrique, CHRU Besançon, Besançon
  - Hôpital de Enfants, Unité Onco-Hématologie Pédiatrique, Groupe Hospitalier Pellegrin, Bordeaux
  - Département de Pédiatrie et Génétique Médicale CHRU Morvan, Brest
  - Unité d'hémato-immuno-oncologie pédiatrique. Centre Hospitalier Universitaire niveau 1 - bâtiment FEH, Caen
  - Unité Onco- Hématologie Pédiatrique CHU Estaing 1 place Lucie-Aubrac, Clermont-Ferrand
  - Service Immuno-Hématologie Oncologie Pédiatrique, Dijon
  - Service onco hématologie pédiatrique CHU de Grenoble site Nord - Hôpital Couple enfant, Grenoble
  - Unité d'hématologie pédiatrique CHRU de Lille - Hôpital Jeanne de Flandre, Lille
  - Service d'Hématologie - Oncologie pédiatrique CHU Limoges - Hôpital de la mère et de l'enfant, Limoges
  - Service d'immuno-hématologie pédiatrique et de transplantation de moelle osseuse, CHU de Lyon HCL - GH Est-Institut d'hématologie et d'oncologie pédiatrique IHOP, Lyon
  - Service de Pédiatrie et hématologie pédiatrique, CHU de Marseille - Hôpital de la Timone, Marseille
  - UAM Hématologie et Oncologie Pédiatrique, CHU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - Service d'hématologie et oncologie pédiatriques, Hôpital enfant-adolescent, CHU NANTES, Nantes
  - Service d'hémato-oncologie pédiatrique CHU NICE - Hôpital l'Archet 2, Nice
  - service d'oncologie pédiatrique, institut Curie, Paris
  - Service Hémato-immuno- oncologie- CHU PARIS Armand Trousseau, Paris
  - Service d' hémato-immunologie CHU Paris - Hôpital Robert Debré, Paris
  - Service Oncologie-Hématologie pédiatrique CHU de Poitiers, Poitiers
  - Service d'Hémato-Oncologie Pédiatrique- American Hospital, Reims
  - Pôle pédiatrie Hémato-cancérologie pédiatrique- CHU RENNES - Hôpital sud, Rennes
  - Service d'Hemato-Oncologie Pediatrique CHU Rouen, Rouen
  - service d'oncologie pédiatrique, hopital Félix Guyon, Saint-Denis
  - Pôle mère enfant-Unité Hématologie - Oncologie pédiatrique - CHU Hôpital NORD, Saint-Priest-en-Jarez
  - Service d'Onco-Hematologie Pediatrique CHU STRASBOURG -Hôpital de Hautepierre, Strasbourg
  - Service Pédiatrie - Hématologie Immunologie Oncologie - CHU Toulouse, Toulouse
  - Service d'hémato-oncologie pédiatrique- CHU de Nancy - Hôpital de Brabois Enfant, Vandœuvre-lès-Nancy
  - Dépt de Pédiatrie Gustave Roussy, Villejuif
- Germany (55):
  - Universitätsklinikum Aachen .Klinik für Kinder - und Jugendmedizin Hämatologie / Onkologie, Aachen
  - Klinikum Augsburg ,Schwäbisches Kinderkrebszentrum. I. Klinik für Kinder und Jugendliche Hämatologie / Onkologie, Augsburg
  - HELIOS Klinikum Berlin-Buch, Kinderklinik, Pädiatrische Hämatologie und Onkologie, Berlin
  - Charité Campus Virchow-Klinikum, Zentrum für Kinder- und Jugendmedizin- Abt. Hämatologie / Onkologie, Berlin
  - Evangelisches Krankenhaus Bielefeld GmbH, Klinik für Kinder- und Jugendmedizin, Hämatologie und Onkologie, Bielefeld
  - Zentrum für Kinderheilkunde der Universität Bonn, Abt. Päd. Hämatologie / Onkologie, Bonn
  - Städtisches Klinikum Braunschweig gGmbH, Zentrum für Kinder- und Jugendmedizin, Braunschweig
  - Klinikum Bremen-Mitte gGmbH, Prof.-Hess-Kinderklinik,Pädiatrische Onkologie und Hämatologie, Bremen
  - Klinikum Chemnitz gGmbH, Klinik für Kinder- und Jugendmedizin, Päd. Hämatologie und Onkologie, Chemnitz
  - Klinikum der Universität zu Köln, Klinik für Kinder- und Jugendmedizin, Abt. Kinderonkologie und -hämatologie, Cologne
  - Carl-Thiem-Klinikum, Kinderklinik, Station 5e, Cottbus
  - Vestische Kinderklinik, Universität Witten / Herdecke, Datteln
  - Klinikum Dortmund gGmbH, Klinik für Kinder- und Jugendmedizin, Station K1, Abt. Päd. Onkologie / Hämatologie, Dortmund
  - Universitätsklinik Carl Gustav Carus der TU Dresden, Klinik für Kinder- und Jugendmedizin, Dresden
  - Universitätsklinikum Düsseldorf, Zentrum für Kinder- und Jugendmedizin, Klinik für Päd. Hämatologie und Onkologie, Düsseldorf
  - HELIOS Klinikum Erfurt GmbH, Klinik für Kinder- und Jugendmedizin, Päd. Onkologie / Hämatologie, Erfurt
  - Universitätsklinikum Erlangen, Klinik für Kinder- und Jugendmedizin, Pädiatrische Onkologie / Hämatologie, Erlangen
  - Universitätsklinikum Essen, Zentrum für Kinder- und Jugendmedizin, Hämatologie / Onkologie, Essen
  - Universitätsklinikum Frankfurt, Klinik für Kinder- und Jugendmedizin, Pädiatrische Hämatologie und Onkologie, Frankfurt
  - Universitätsklinikum Freiburg, Zentrum für Kinder- und Jugendmedizin, Klinik IV: Päd. Hämatologie und Onkologie, Freiburg im Breisgau
  - Universitätsklinikum Gießen und Marburg, Standort Gießen, Zentrum für Kinderhämatologie und -onkologie, Giessen
  - Georg-August-Universität Universitäts-Kinderklinik, Pädiatrie I, Göttingen
  - Universitätsklinikum Greifswald KdöR, Klinik und Poliklinik für Kinder- und Jugendmedizin, Abt. Pädiatrische Onkologie und Hämatologie, Greifswald
  - Universitätsklinikum Halle (Saale), Klinik für Kinder- und Jugendmedizin, Pädiatrische Hämatologie / Onkologie, Halle
  - Universitätsklinikum Hamburg Eppendorf, Zentrum für Kinder- und Jugendmedizin, Abt. Pädiatrische Hämatologie und Onkologie, Hamburg
  - Medizinische Hochschule Hannover, Kinderheilkunde, Päd. Hämatologie / Onkologie, Hanover
  - Universitäts-Kinderklinik Heidelberg, Abt. Hämatologie / Onkologie, Heidelberg
  - Gemeinschaftskrankenhaus Herdecke, Kinder- und Jugendmedizin, Päd. Hämatologie / Onkologie, Herdecke
  - Universitätskliniken für Kinder- und Jugendmedizin, Päd. Hämatologie und Onkologie, Geb. 9, Homburg
  - Universitätsklinikum Jena, Klinik für Kinder- und Jugendmedizin, Jena
  - Städtisches Klinikum Karlsruhe gGmbH, Kinderklinik, Station S 24, Karlsruhe
  - Klinikum Kassel Gesundheit Nordhessen Holding AG, Klinik für pädiatrische Hämatologie und Onkologie, Kassel
  - Universitätsklinikum Schleswig Holstein Campus Kiel, Klinik für Allgemeine Pädiatrie, Päd. Onkologie / Hämatologie, Kiel
  - Gemeinschaftsklinikum Mittelrhein Kemperhof, Klinik für Kinder- und Jugendmedizin, Pädiatrische Hämatologie und Onkologie, Koblenz
  - HELIOS Klinikum Krefeld, Zentrum für Kinder- und Jugendmedizin, Päd. Hämatologie/Onkologie, Krefeld
  - Universitätsklinikum Leipzig, Klinik für Kinder und Jugendliche, Abt. Päd. Hämatologie / Onkologie, Leipzig
  - Universitätsklinikum Schleswig Holstein Campus Lübeck, Klinik für Kinder- und Jugendmedizin, Hämatologie und Onkologie, Lübeck
  - Universitätsklinikum Magdeburg A. ö. R., Kinderklinik, Päd. Hämatologie / Onkologie, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Zentrum für Kinder- und Jugendmedizin, Pädiatrische Hämatologie / Onkologie, Mainz
  - Klinikum Mannheim gGmbH, Universitäts-Kinderklinik, Päd. Onkologie /Hämatologie, Manheim
  - Johannes Wesling Klinikum Minden, Klinik für Kinder- und Jugendmedizin, Päd. Hämatologie / Onkologie, Station E 22, Minden
  - Klinikum der LMU, Dr. von Haunersches Kinderspital, Pädiatrische Hämatologie / Onkologie, München
  - Klinikum Schwabing, Kinderklinik der TU Päd. Hämatologie / Onkologie, Station 24d, München
  - Universitätsklinikum Münster, Klinik für Kinder- und Jugendmedizin, Abt. Pädiatrische Hämatologie und Onkologie, Münster
  - Diakonie Neuendettelsau, Kliniken Hallerwiese / Cnopf'sche Kinderklinik, Pädiatrische Hämatologie /Onkologie, Nuremberg
  - Klinikum Oldenburg AöR, Zentrum für Kinder- und Jugendmedizin, Abt. Hämatologie / Onkologie, Oldenburg
  - Universitätsklinikum Regensburg, Klinik für Kinder- und Jugendmedizin, Abt. Päd. Hämatologie, Onkologie, SZT, Regensburg
  - Universitätsklinikum Rostock, Kinder- und Jugendklinik, Päd. Hämatologie und Onkologie, Rostock
  - Asklepios Klinik St. Augustin GmbH, Kinder- und Jugendmedizin, Kinder-Hämatologie und Onkologie, Sankt Augustin
  - HELIOS Kliniken Schwerin GmbH, Klinik für Kinder- und Jugendmedizin, Station A1, Schwerin
  - Klinikum Stuttgart, Olgahospital Zentrum für Kinder- und Jugendmedizin Pädiatrie 5 (Onkologie, Hämatologie, Immunologie), Stuttgart
  - Klinikum Mutterhaus der Borromäerinnen gGmbH, Pädiatrische Abteilung, Trier
  - Universitätsklinik Tübingen, Klinik für Kinderheilkunde und Jugendmedizin, Päd. Hämatologie / Onkologie, Tübingen
  - Universitätsklinikum Ulm, Klinik für Kinder- und Jugendmedizin, Päd. Hämatologie und Onkologie, Ulm
  - Universitätskinderklinik Würzburg, Päd. Onkologie und Hämatologie, Würzburg
- Hungary (6):
  - 2nd Dep. of Pediatrics, Semmelweis Univ, Budapest
  - Heim Pal Children Hospital, Budapest
  - Dep. of Pediatrics, Univ. of Debrecen, Debrecen
  - Children's Treating Center, Miskolc, Miskolc
  - Dep. of Pediatrics, University of Pecs, Pécs
  - Dep. of Pediatrics, Univ. of Szeged, Szeged
- Our Lady's Children's Hospital Crumlin, Dublin, Ireland
- Israel (6):
  - Children's Hospital at Soroka Medical Center, Beersheba
  - Ruth Rappaport Children's Hospital, Rambam Medical Center, Haifa
  - Children's Hospital at Hadassah, Ein Kerem Medical Center, Jerusalem
  - Schneider Children's hospital, Rabin Medical Center, Petah Tikva
  - Edmond and Lily Safra Children's Hospital, Sheba Medical Center, Ramat Gan
  - Dana Children's Hospital, Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (33):
  - Azienda Ospedaliero Universitaria Delle Marche, Ancona
  - University Hospital Consorziale Policlinico, Bari
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliero-Universitaria Di Bologna IRCCS, Bologna
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia
  - ARNAS G. Brotzu, Cagliari
  - Azienda Ospedaliero Universitaria Policlinico G Rodolico San Marco Di Catania, Catania
  - University Hospital Of Ferrara, Cona
  - U. O. di Pediatria- Azienda Ospedaliera Annunziata, Cosenza
  - Dipartimento di Medicina Clinica e Sperimentale Sezione di Pediatria - Università di Ferrara, Ferrara
  - Azienda Ospedaliera Universitaria Meyer IRCCS, Florence
  - Giannina Gaslini Institute For Scientific Hospitalization And Care, Genova
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliero Universitaria di Modena, Modena
  - Fondazione IRCCS San Gerardo Dei Tintori, Monza
  - L'Azienda Ospedaliera Di Rilievo Nazionale Santobono-Pausilipon, Naples
  - S.C. Ematologia Oncologica- Ospedale "Pausilipon", Napoli
  - Azienda Ospedale-Università Padova, Padua
  - ARNAS Civico Di Cristina Benfratelli, Palermo
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Perugia
  - Azienda Sanitaria Locale Di Pescara, Pescara
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Unità Sanitaria della Romagna, Rimini
  - Sezione Ematologia- Dipart. Biotecnico Cellulare ed Ematologia- Università "La Sapienza", Roma
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Casa Sollievo Della Sofferenza, San Giovanni Rotondo
  - Oncologia Pediatrica,- Ospedale "R. Silvestrini", San Sisto
  - Azienda Ospedaliera Universitaria Città Della Salute E Della Scienza Di Torino, Torino
  - Istituto Di Ricovero E Cura A Carattere Scientifico Materno Infantile Burlo Garofolo, Trieste
  - Azienda Socio Sanitaria Territoriale Dei Sette Laghi, Varese
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona
- Princess Maxima Centre for Pediatric Oncology, Utrecht, Netherlands
- Norway (3):
  - Haukeland University Hospital in Bergen, Bergen
  - University Hospital Northern Norway, Tromsø
  - St Olavs Hospital in Trondheim, Trondheim
- Poland (16):
  - Department of Pediatric Oncology and Hematology, Medical University of Bialystok, Bialystok
  - Department of Pediatric Hematology and Oncology, Nicolaus Copernicus University, Bydgoszcz
  - Department of Pediatric Hematology and Oncology, Center of Pediatrics and Oncology in Chorzów, Chorzów
  - Department of Pediatrics, Hematology, Oncology and Endocrinology, Medical University of Gdansk, Gdansk
  - Department of Pediatric Oncology and Hematology, Center of Pediatrics in Kielce, Kielce
  - Department of Pediatric Oncology/Hematology, Institute of Pediatrics, Medical College Jagiellonian University, Krakow
  - Department of Pediatrics, Oncology, Hematology and Diabetology, Institute of Pediatrics, Medical University of Lodz, Lodz
  - Department of Pediatric Hematology, Oncology and Transplantology, Medical University of Lublin, Lublin
  - Department of Pediatric Oncology and Hematology, Provincial Specialist Children's Hospital, Olsztyn
  - Department of Pediatric Oncology, Hematology and Transplantology, Poznan University of Medical Sciences, Poznan
  - Department of Paediatric Oncology and Haematology, University of Rzeszów, Department of Pediatrics, Rzeszów
  - Department of Pediatrics, Children Hematology nad Oncology, Pomeranian Medical University, Szczecin
  - Department of Pediatrics, Hematology and Oncology, Medical University of Warsaw, Warsaw
  - Department of Pediatric Oncology, Children's Memorial Health Institute, Warsaw
  - Department of Bone Marrow Transplantation, Children Oncology and Hematology, Wroclaw Medical University, Wroclaw
  - Department of Pediatric Hematology and Oncology, Silesian Medical University in Katowice, Zabrze
- Portugal (3):
  - Centro Hospitalar e Universitário de Coimbra, Coimbra
  - Instituto Português de Oncologia - Francisco Gentil - Libosa, Lisbon
  - Instituto Português de Oncologia - Francisco Gentil - Porto, Porto
- Russia (2):
  - National Center for Pediatric Hematology, Oncology and Immunology Moscow, Moscow
  - Oncological center of regional Children's Hospital, Yekaterinburg
- Slovakia (3):
  - Department of pediatric oncology and hematology, Children´s Faculty Hospital, Banská Bystrica
  - Department of pediatric hematology and oncology, National Institute of Children's Diseases, Bratislava
  - Department of pediatric hematology and oncology, Children´s University Hospital, Košice
- Spain (30):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Torrecárdenas, Almería
  - Hospital Materno-Infantil de Badajoz, Badajoz
  - Hospital Universitario Cruces, Barakaldo
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Sant Joan de Déu, Esplugues de Llobregat
  - Hospital Universitario Virgen de las Nieves, Granada
  - Complejo Hospitalario Universitario Insular Materno Infantil, Las Palmas de Gran Canaria
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Virgen del Camino, Pamplona
  - Complejo Hospitalario Universitario de Vigo, Pontevedra
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (6):
  - Barncancercentrum, Drottning Silvias Barn och Ungdomssjukhus, Sahlgrenska Universitetssjukhuset, Gothenburg
  - Barnonkologiska enheten, Barn och Ungdomsmedicinska kliniken, Universitetssjukhuset i Linköping, Linköping
  - Barnonkologi, Skåne Universitetssjukhus, Lund
  - Barncanceravdelningen Astrid Lindgrens Barnsjukhus, Nya Karolinska Universitetssjukhuset, Stockholm
  - Barnonkologiska avdelningen, Barn 3, Norrlands Universitetssjukhus, Umeå
  - Barnavdelningen för blod- och tumörsjukdomar 95A, Akademiska sjukhuset, Uppsala
- Switzerland (9):
  - Kantonsspital Aarau, Aarau
  - Universitäts-Kinderspital beider Basel (UKBB), Basel
  - Ospedale San Giovanni, Bellinzona
  - Inselspital Bern, University of Bern, Bern
  - HUG Hôpitaux Universitaires de Genève, Geneva
  - CHUV - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Luzerner Kantonspital - Kinderspital Luzern, Lucerne
  - Ostschweizer Kinderspital, Sankt Gallen
  - Universitäts-Kinderspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khanam T, Sandmann S, Seggewiss J, Ruether C, Zimmermann M, Norvil AB, Bartenhagen C, Randau G, Mueller S, Herbrueggen H, Hoffmann P, Herms S, Wei L, Woeste M, Wuensch C, Gowher H, Oschlies I, Klapper W, Woessmann W, Dugas M, Burkhardt B. Integrative genomic analysis of pediatric T-cell lymphoblastic lymphoma reveals candidates of clinical significance. Blood. 2021 Apr 29;137(17):2347-2359. doi: 10.1182/blood.2020005381. PMID 33152759